CLINICAL TRIAL: NCT02992899
Title: Closed Loop Vagal Nerve Stimulation in Patients With Posttraumatic Stress Disorder
Brief Title: Closed Loop Vagal Nerve Stimulation for Patients With Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Institute of Technology (Other)
Responsible Party: Principal Investigator, J. Douglas Bremner, MD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00091171
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Results first posted 2021-05-19 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: PostTraumatic Stress Disorder
Keywords: stress disorders, post-traumatic; posttraumatic stress disorder; PTSD; vagal nerve
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Vagal Nerve Stimulation (Experimental): Participants randomized to this arm will receive stimulation of the vagus nerve in conjunction with stress exposure.
  Interventions: Device: GammaCore/electroCore non-invasive VNS device; Drug: O-15 water
- Sham Stimulation (Sham Comparator): Participants randomized to this arm will receive sham stimulation of the vagus nerve in conjunction with stress exposure.
  Interventions: Device: Sham gammaCore/electroCore; Drug: O-15 water

INTERVENTIONS:
Device: GammaCore/electroCore non-invasive VNS device — Vasal nerve stimulation (VNS) is self-administered using the electroCore non-invasive VNS device. The intensity of the stimulus (the current amplitude) is adjusted by the user, to the maximum tolerable level to ensure VNS without causing excessive pain (typically 10-30 V), the burst frequency to 5 kilohertz (kHz), and the envelope frequency to 25 Hz. These are the standard frequency settings that electroCore has demonstrated to be most effective in capturing the vagus nerve based on evoked potential studies. The duration of delivery is 2 minutes, one minute into which the high-resolution positron emission tomography (HR-PET) scan is conducted; following an additional 8 minutes, a second VNS delivery is administered, after which another scan is obtained.
  Arms: Vagal Nerve Stimulation
Device: Sham gammaCore/electroCore — Sham vasal nerve stimulation (VNS) is self-administered using the electroCore non-invasive VNS device. The device is programmed such that no actual stimulation is given to the vagus nerve. The duration of delivery is 2 minutes, one minute into which the HR-PET scan is conducted; following an additional 8 minutes, a second sham VNS delivery is administered, after which another scan is obtained.
  Arms: Sham Stimulation
Drug: O-15 water — Oxygen-15 labelled water is a radioactive variation of regular water, in which the oxygen atom has been replaced by oxygen-15 (15O), a positron-emitting isotope. 15O-water is used as a radioactive tracer for measuring and quantifying blood flow using positron emission tomography (PET) . H2[15O] will be prepared on-site in the Emory PET Center cyclotron. During the hours of the test, an intravenous infusion of normal saline will be started to permit the bolus injection of H2[15O]. Subjects will receive a 20 mCi intravenous bolus of H2[15O] for each of the 14 scans during exposure to neutral and traumatic scripts.

SUMMARY:
The tasks of the project are to map the potency and kinetics of the neurologic, autonomic peripheral, inflammatory, and behavioral responses to vagal nerve stimulation (VNS) vs. sham treatment, at baseline and in response to stressful traumatic scripts related to personal traumatic events, as well as a series of other stressors.

DETAILED DESCRIPTION:
The purpose of this project is to develop the fundamental physiological understanding of feedback controlled vagal nerve stimulation (VNS) using positron emission tomography (PET) brain imaging and blood biomarker measurement with stress in healthy individuals and individuals with PTSD. Healthy human subjects with a history of psychological trauma but without the diagnosis of a psychiatric disorder (Phase 1), and human subjects with a history of PTSD (Phase 2), undergo PET imaging of the brain in conjunction with VNS or a sham treatment during exposure to neutral scripts and scripts of personal traumatic events. Blood is drawn simultaneously for measurement of a variety of stress responsive biomarkers, including inflammatory markers and neurohormones. A second PET scan with biomarkers assesses the delayed effects of VNS. On two other days subjects undergo exposure to random stressors with VNS or sham in conjunction with measurement of stress biomarkers.

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

* Do not meet criteria for post traumatic stress disorder (PTSD) or other major mental disorder as determined by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5 SCID) interview for PTSD
* Have a history of psychological trauma as defined by DSM-5.

Phase 2:

- Meet criteria for PTSD as determined by the Structured Clinical Interview for DSM-5 (SCID) interview for PTSD.

Exclusion Criteria:

* Positive pregnancy test
* Meningitis
* Traumatic brain injury
* Neurological disorder or organic mental disorder
* History of loss of consciousness greater than one minute
* Alcohol abuse or substance abuse or dependence based on the SCID within the past 12 months
* Positive toxicology screen
* Current or lifetime history of schizophrenia, schizoaffective disorder, or bulimia, based on the SCID
* A history of serious medical or neurological illness, such as cardiovascular, gastrointestinal, hepatic, renal, neurologic or other systemic illness
* Evidence of a major medical or neurological illness on physical examination or as a result of laboratory studies (complete blood count (CBC), blood urea nitrogen (BUN), creatinine, blood sugar, electrolytes, liver and thyroid function tests, urinalysis, and EKG)
* Active implantable device (i.e. pacemaker)
* Carotid atherosclerosis
* Cervical vagotomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2019-09-21 (Actual); Study Completion 2019-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Bremner, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wittbrodt MT, Gurel NZ, Nye JA, Shandhi MMH, Gazi AH, Shah AJ, Pearce BD, Murrah N, Ko YA, Shallenberger LH, Vaccarino V, Inan OT, Bremner JD. Noninvasive Cervical Vagal Nerve Stimulation Alters Brain Activity During Traumatic Stress in Individuals With Posttraumatic Stress Disorder. Psychosom Med. 2021 Nov-Dec 01;83(9):969-977. doi: 10.1097/PSY.0000000000000987. PMID 34292205
- [Derived] Gurel NZ, Wittbrodt MT, Jung H, Shandhi MMH, Driggers EG, Ladd SL, Huang M, Ko YA, Shallenberger L, Beckwith J, Nye JA, Pearce BD, Vaccarino V, Shah AJ, Inan OT, Bremner JD. Transcutaneous cervical vagal nerve stimulation reduces sympathetic responses to stress in posttraumatic stress disorder: A double-blind, randomized, sham controlled trial. Neurobiol Stress. 2020 Oct 20;13:100264. doi: 10.1016/j.ynstr.2020.100264. eCollection 2020 Nov. PMID 33344717
- [Derived] Gazi AH, Gurel NZ, Richardson KLS, Wittbrodt MT, Shah AJ, Vaccarino V, Bremner JD, Inan OT. Digital Cardiovascular Biomarker Responses to Transcutaneous Cervical Vagus Nerve Stimulation: State-Space Modeling, Prediction, and Simulation. JMIR Mhealth Uhealth. 2020 Sep 22;8(9):e20488. doi: 10.2196/20488. PMID 32960179

RESULTS

PARTICIPANT FLOW:
Groups:
- Vagal Nerve Stimulation: Participants randomized to this arm will receive stimulation of the vagus nerve in conjunction with stress exposure.
  GammaCore/electroCore non-invasive VNS device: Vasal nerve stimulation (VNS) is self-administered using the electroCore non-invasive VNS device. The intensity of the stimulus is adjusted by the user, to the maximum tolerable level to ensure VNS without causing excessive pain (typically 10-30 V). The duration of delivery is 2 minutes, one minute into which the high-resolution positron emission tomography (HR-PET) scan is conducted; following an additional 8 minutes, a second VNS delivery is administered, after which another scan is obtained.
  O-15 water: Oxygen-15 labelled water is a radioactive variation of regular water, in which the oxygen atom has been replaced by oxygen-15 (15O), a positron-emitting isotope. 15O-water is used as a radioactive tracer for measuring and quantifying blood flow using positron emission tomography (PET) . Subjects will receive a 20 mCi intravenous bolus of H2[15O] for each of the 14 scans during exposure to neutral and traumatic scripts.
Period: Overall Study
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Started | 27 | 29
Completed | 25 | 26
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation | Total
Number analyzed (Participants) | 27 | 29 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (11) | 35 (11) | 33 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 11 | 13 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 13 | 14 | 27
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 27 | 29 | 56

OUTCOME MEASURES:

1. Primary Outcome: Level of Interleukin-6 (IL6)
Description: IL6 level will be collected via blood draw. Change is defined as the difference in IL6 level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: Due to technical reasons and/or limited blood draw, the number of participants analyzed is less than the number of participants that completed the trial.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 23 | 22
pg/ml
  Baseline IL-6 Level | 0.88 (0.59) | 0.84 (0.61)
  Post Stress Testing IL-6 Level | 1.77 (1.43) | 2.11 (2.49)

2. Secondary Outcome: Level of Tryptophan
Description: Tryptophan level will be collected via blood draw. Change is defined as the difference in tryptophan level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micromole/l
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 16 | 17
micromole/l
  Baseline Tryptophan Level | 50.59 (11.65) | 55.80 (15.74)
  Post Stress Testing Tryptophan Level | 54.42 (13.21) | 57.79 (14.38)

3. Secondary Outcome: Level of Kynurenine
Description: Kynurenine level will be collected via blood draw. Change is defined as the difference in kynurenine level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 16 | 18
µM
  Baseline Kynurenine Level | 4.72 (5.37) | 7.19 (5.01)
  Post Stress Testing Kynurenine Level | 5.04 (5.81) | 7.06 (5.64)

4. Secondary Outcome: Level of Kynurenic Acid
Description: Kynurenic acid level will be collected via blood draw. Change is defined as the difference in kynurenic acid level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/100 microliters
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 7 | 11
pmol/100 microliters
  Baseline Kynurenic Acid Level | 35.71 (9.59) | 43.07 (21.13)
  Post Stress Testing Kynurenic Acid Level | 38.81 (16.50) | 37.88 (12.37)

5. Secondary Outcome: Level of 3-3 Hydroxykynurenine
Description: 3-3 hydroxykynurenine level will be collected via blood draw. Change is defined as the difference in 3-3 hydroxykynurenine level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: This outcome was not assessed due to a lack of resources and a focus on other pertinent biomarkers per the literature.
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Level of Anthranilic Acid
Description: Anthranilic Acid level will be collected via blood draw. Change is defined as the difference in anthranilic acid level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 16 | 17
nM
  Baseline Anthranilic Acid Level | 8.32 (2.68) | 7.02 (1.68)
  Post Stress Testing Anthranilic Acid Level | 7.49 (2.13) | 6.90 (1.59)

7. Secondary Outcome: Level of Tumor Necrosis Factor (TNF)-Alpha
Description: TNF-alpha level will be collected via blood draw. Change is defined as the difference in TNF-alpha level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 16 | 14
pg/mL
  Baseline Tumor Necrosis Factor (TNF)-alpha Level | 2.81 (1.28) | 2.37 (0.87)
  Post Stress Testing Tumor Necrosis Factor (TNF)-alpha Level | 2.63 (1.03) | 2.26 (0.74)

8. Secondary Outcome: Level of Interferon-Gamma
Description: Interferon-Gamma level will be collected via blood draw. Change is defined as the difference in Interferon-Gamma level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 23 | 22
pg/mL
  Baseline Interferon-Gamma Level | 4.75 (9.61) | 3.43 (2.58)
  Post Stress Testing Interferon-Gamma Level | 4.86 (10.20) | 8.87 (27.33)

9. Secondary Outcome: Level of Interleukin-1 Beta
Description: Interleukin-1 Beta level will be collected via blood draw. Change is defined as the difference in Interleukin-1 Beta level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 16 | 14
pg/mL
  Baseline Interleukin-1 Beta Level | 0.056 (0.033) | 0.086 (0.056)
  Post Stress Testing Interleukin-1 Beta Level | 0.071 (0.041) | 0.085 (0.077)

10. Secondary Outcome: Level of Interleukin-2 (IL2)
Description: IL2 level will be collected via blood draw. Change is defined as the difference in IL2 level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 16 | 14
pg/ml
  Baseline Interleukin-2 (IL2) Level | 0.29 (0.22) | 0.29 (0.20)
  Post Stress Testing Interleukin-2 (IL2) Level | 0.36 (0.20) | 0.27 (0.20)

11. Secondary Outcome: Level of Interleukin-4 (IL4)
Description: IL4 level will be collected via blood draw. Change is defined as the difference in IL4 level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: This outcome was not assessed due to a lack of resources and a focus on other pertinent biomarkers per the literature.
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Level of Interleukin-8 (IL8)
Description: IL8 level will be collected via blood draw. Change is defined as the difference in IL8 level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: This outcome was not assessed due to a lack of resources and a focus on other pertinent biomarkers per the literature.
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Level of Interleukin-10 (IL10)
Description: IL10 level will be collected via blood draw. Change is defined as the difference in IL10 level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: This outcome was not assessed due to a lack of resources and a focus on other pertinent biomarkers per the literature.
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Level of Interleukin-12p70 (IL12p70)
Description: IL12p70 level will be collected via blood draw. Change is defined as the difference in IL12p70 level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 21 | 20
pg/ml
  Baseline Interleukin-12p70 (IL12p70) Level Level | 2.20 (1.48) | 3.22 (1.68)
  Post Stress Testing Interleukin-12p70 (IL12p70) Level Level | 1.82 (0.99) | 2.96 (2.02)

15. Secondary Outcome: Level of Interleukin-12p (IL12p)
Description: IL12p level will be collected via blood draw. Change is defined as the difference in IL12p level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: This outcome was not assessed due to a lack of resources and a focus on other pertinent biomarkers per the literature.
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Level of Interleukin-13 (IL13)
Description: IL13 level will be collected via blood draw. Change is defined as the difference in IL13 level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 21 | 20
pg/ml
  Baseline Interleukin-13 (IL13) Level | 33.77 (16.87) | 43.10 (18.78)
  Post Stress Testing Interleukin-13 (IL13) Level | 29.17 (14.03) | 43.55 (31.91)

17. Secondary Outcome: Level of Macrophage Migration Inhibitory Factor
Description: Macrophage migration inhibitory factor will be collected via blood draw. Change is defined as the difference in factor level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 21 | 20
pg/ml
  Baseline Macrophage Migration Inhibitory Factor Level | 32,204 (14,130) | 31,309 (20,624)
  Post Stress Testing Macrophage Migration Inhibitory Factor Level | 30,403 (14,007) | 30,515 (17,399)

18. Secondary Outcome: Level of High-Mobility Group Protein B1
Description: High-mobility group protein B1 level will be collected via blood draw. Change is defined as the difference in high-mobility group protein B1 level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 22 | 21
ng/mL
  Baseline High-Mobility Group Protein B1 Level | 1,552 (1,105) | 1,734 (893)
  Post Stress Testing High-Mobility Group Protein B1 Level | 1,299 (574) | 1,691 (942)

19. Secondary Outcome: Level of Adrenocorticotropic Hormone
Description: Adrenocorticotropic hormone level will be collected via blood draw. Change is defined as the difference in adrenocorticotropic hormone level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: This outcome was not assessed due to a lack of resources and a focus on other pertinent biomarkers per the literature.
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Level of Cortisol
Description: Cortisol level will be collected via blood draw. Change is defined as the difference in cortisol level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: This outcome was not assessed due to a lack of resources and a focus on other pertinent biomarkers per the literature.
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Level of Epinephrine
Description: Epinephrine level will be collected via blood draw. Change is defined as the difference in epinephrine level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: This outcome was not assessed due to a lack of resources and a focus on other pertinent biomarkers per the literature.
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Level of Dopamine
Description: Dopamine level will be collected via blood draw. Change is defined as the difference in dopamine level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: This outcome was not assessed due to a lack of resources and a focus on other pertinent biomarkers per the literature.
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Level of Norepinephrine
Description: Norepinephrine level will be collected via blood draw. Change is defined as the difference in norepinephrine level from baseline to post emotional stress testing.
Time Frame: Baseline, Post Stress Testing (Up to 4 Hours)
Population: This outcome was not assessed due to a lack of resources and a focus on other pertinent biomarkers per the literature.
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time consent was given through all follow up (up to 4 hours post intervention).
Arm/Group | Vagal Nerve Stimulation | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/29
Other Adverse Events (participants affected / at risk) | 0/27 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT02992899/Prot_SAP_000.pdf